CLINICAL TRIAL: NCT04620109
Title: A Phase 1 Randomized, Double Blinded, Placebo-Controlled Single Dose and Repeat Dose Escalation Study to Evaluate Safety and Tolerability and Pharmacokinetic Characteristics of KDR2-2 in Adult Healthy Male and Female Volunteers
Brief Title: Clinical Evaluation of Safety and Tolerability of KDR2-2 Eye Drops in Healthy Volunteers With Pharmacokinetic Assessment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou HuiBoRui Biological Pharmaceutical Technology Co. Ltd (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HBR2019-101
Record Dates: First submitted 2020-10-19; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Corneal Neovascularization
Keywords: Corneal neovascularization
MeSH Terms: conditions — Corneal Neovascularization

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- SDE Placebo (Placebo Comparator): Subjects will receive placebo (drops without drug).
  Interventions: Drug: Placebo
- SDE 0.03 mg/eye (Active Comparator): Actual dose is 0.03 mg/eye by 60μL KDR2-2 eyedrops of a concentration of 0.5 mg/mL for 1 time.
  Interventions: Drug: KDR2-2
- SDE 0.06 mg/eye (Active Comparator): Actual dose is 0.06 mg/eye by 60μL KDR2-2 eyedrops of a concentration of 1.0 mg/mL for 1 time.
  Interventions: Drug: KDR2-2
- SDE 0.12 mg/eye (Active Comparator): Actual dose is 0.12 mg/eye by 60μL KDR2-2 eyedrops of a concentration of 2.0 mg/mL for 1 time.
  Interventions: Drug: KDR2-2
- SDE 0.24 mg/eye (Active Comparator): Actual dose is 0.24 mg/eye by 60μL KDR2-2 eyedrops of a concentration of 4 mg/mL for 1 time.
  Interventions: Drug: KDR2-2
- RDE 0.06 mg/eye (Active Comparator): The actual dosage is 0.06 mg/eye given 4 times a day for a maximum daily dosage of 0.24mg (60μL KDR2-2 eyedrops concentration of 1.0 mg/mL), which will continues for 6 days plus 1 administration of 0.06 mg/eye in the morning of Day 7. That cohort only started after safety proof from SDE 0.24 mg/eye cohort.
  Interventions: Drug: KDR2-2
- RDE 0.12 mg/eye (Active Comparator): The actual dosage is 0.12 mg/eye given 4 times a day for a maximum daily dosage of 0.48mg (60μL KDR2-2 eyedrops concentration of 2.0 mg/mL), which will continues for 6 days plus 1 administration of 0.12 mg/eye in the morning of Day 7. That cohort might be optional based on emerging data from this study.
  Interventions: Drug: KDR2-2
- RDE 0.24 mg/eye (Active Comparator): The actual dosage is 0.24 mg/eye given 4 times a day for a maximum daily dosage of 0.96mg (60μL KDR2-2 eyedrops concentration of 4.0 mg/mL), which will continues for 6 days plus 1 administration of 0.24 mg/eye in the morning of Day 7. That cohort might be optional based on emerging data from this study.
  Interventions: Drug: KDR2-2
- RDE Placebo (Placebo Comparator): Subjects will receive placebo (drops without drug).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KDR2-2 — KDR2-2 is a synthetic anti-angiogenic chemical compound with highly effective inhibition on vascular endothelial growth factor receptor-2 (VEGFR2), and an additional, moderate inhibitory effect on platelet-derived growth factor receptor β (PDGFRβ).
  KDR2-2 suspension eye drop is in development for the treatment of corneal neovascularization.
  Other Names: KDR2-2 suspension eyedrop; KDR2-2 ophthalmic suspension
  Arms: RDE 0.06 mg/eye; RDE 0.12 mg/eye; RDE 0.24 mg/eye; SDE 0.03 mg/eye; SDE 0.06 mg/eye; SDE 0.12 mg/eye; SDE 0.24 mg/eye
Drug: Placebo — Placebo : the formulation and the product process of placebo are the same as the KDR2-2 eye drops, but without API .
  Arms: RDE Placebo; SDE Placebo

SUMMARY:
A Phase 1 randomized, double blinded, placebo-controlled, single dose escalation (SDE) and repeat dose escalation (RDE) study to evaluate safety and tolerability, and PK of KDR2-2 in healthy volunteers. The planned single dose levels are 0.03, 0.06, 0.12, and 0.24 mg/eye, and repeat dose levels are 0.06, 0.12, and 0.24 mg/eye, QID, × 6 days (one dose in the morning on Day 7). Subjects are randomized to KDR2-2 or placebo dosing (6:2 for SDE, or 8:2 for RDE) in each cohorts of relative dosing levels.

DETAILED DESCRIPTION:
This is a Phase 1 randomized, double blinded, placebo-controlled, single dose and repeat dose escalation study to evaluate safety and tolerability, and PK of KDR2-2 in healthy volunteers.

The trial will include a screening period, a treatment period, and a follow-up period of 7 days for single dose escalation (SDE) or repeat dose escalation (RDE) after last administration. The screening period will be up to 28 days prior to investigational product administration. The screening process will initiate upon completion of the informed consent process. Once consent is provided by each participant, a thorough screening process will take place, including detailed medical history, physical examination and ophthalmology examination, vital signs, concomitant medications, safety labs, 12 lead electrocardiogram, serum pregnancy test, urinalysis, serology panel, assessment of inclusion and exclusion criteria. Upon completion of the screening, qualified subjects will be randomized to KDR2-2 or placebo (6:2 for SDE, or 8:2 for RDE). Each enrolled subject will receive one single or repeat assigned dose of KDR2-2 or placebo. The investigator and subjects will be blinded to treatment assignment. During the study, subjects will be evaluated for safety and tolerability, and PK of KDR2-2. In each cohort, a sentinel group of two subjects will be dosed first: one sentinel with KDR2-2, and the other with the placebo. The remaining subjects of the same cohort will be dosed at least 24 hours after sentinel dosing with approval from the principal investigator upon assessing the sentinel group.

KDR2-2 or placebo will be topically administered in the right eye as a single or repeat instillation on Day 1. Subjects will have end-of-study (EOS) follow-up visits on Day 8 (±1) for SDE or Day 15 (±1) for RDE.

The planned single dose levels are 0.03, 0.06, 0.12, and 0.24 mg/eye, and repeat dose levels are 0.06, 0.12, and 0.24 mg/eye, QID, × 6 days (one dose in the morning on Day 7). The Starting dose of KDR2-2 in repeat dose escalation stage will be at least 2 dose levels below the highest single dose level shown to be safe, for example, if 0.24 mg is proven to be safe during SDE, the starting dose during RDE will be 0.06 mg. Other higher dose level(s) might be optional based on emerging data from this study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be enrolled in the trial:

1. Able to understand and willing to sign the ICF
2. Healthy male and female subjects, non-smokers, 18-55 years of age
3. With no significant medical history, and in good health as determined by detailed medical history (neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease), full physical examination, vital signs, 12-lead electrocardiogram (ECG), urinalysis and laboratory tests at screening. For eligibility purposes, abnormal laboratory or vital signs results may be repeated once if abnormal result is observed at the initial reading. Moreover, abnormalities found in the ECG may need to be confirmed by repeated measurements.
4. Subjects must have adequate organ function according to the following laboratory values at Screening and on Day-1. Repeat testing is allowed for verification, at the discretion of the Investigator:

   * Bone marrow function (absolute neutrophil count ≥ 1500/mm3 and platelet count ≥ 100,000/mm3)
   * Adequate liver function [alanine aminotransferase (ALT) ≤ 1.5 × upper limit normal (ULN) and alkaline phosphatase ≤ 1.5 × ULN, total bilirubin ≤ 1.5 mg/dL]
   * Adequate renal function creatinine clearance 60 mL/min based on Cockcroft - Gault equation, or serum creatinine level ≤ 1.5 times the ULN.
5. Be a female of non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is 2 years post-menopausal and have an FSH > 40 mIU/mL, or surgically sterile [defined as having a bilateral oophorectomy, hysterectomy or tubal ligation]) or agree to one of the following to prevent pregnancy and, if a woman of childbearing potential, have a negative serum pregnancy test at screening:

   * If a sexually active woman of childbearing potential (sexually active with a non-sterile male partner) agrees to prevent pregnancy by using double methods of contraception as follow until at least 30 days after the administration of the investigational product:

     1. simultaneous use of intra-uterine contraceptive device, placed at least 4 weeks prior to study drug administration, and condom for the male partner;
     2. simultaneous use of hormonal contraceptives, starting at least 4 weeks prior to study drug administration and must agree to use the same hormonal contraceptive throughout the study, and condom for the male partner;
     3. simultaneous use of diaphragm with intravaginally applied spermicide and male condom for the male partner, starting at least 7 days prior to study drug administration.
   * Male subjects who are not vasectomized for at least 6 months and who are sexually active with a non-sterile female partner must agree to use double methods of contraception below from the first dose of randomized study drug until 7 days after their dose and must not donate sperm during their study participation period:

     1. simultaneous use of a male condom and, for the female partner, hormonal contraceptives (used since at least 4 weeks) or intra-uterine contraceptive device (placed since at least 4 weeks);
     2. simultaneous use of a male condom and, for the female partner, a diaphragm with intravaginally applied spermicide.
6. Body mass index (BMI) 19.0-32.0 kg/m2 and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females.
7. Blood pressure ≤ 139/89 mm Hg at screening and on Day -1. If abnormal findings deemed by the Investigator as not clinically significant, it may be repeated.
8. Subjects are able to follow the study protocol and complete the trial.

Exclusion Criteria:

Subjects who meet any of the following criteria cannot be enrolled:

1. History of severe infection within 4 weeks prior to administration; signs and symptoms of any active infection regardless of severity within 2 weeks prior to administration.
2. History of eye infection, or trauma or surgeries including LASIK.
3. Subjects with a single eye.
4. History of hypersensitivity to similar drugs to KDR2-2 or their excipients.
5. Clinically significant abnormalities on ocular examination, including slit lamp, that would hinder the assessment of the eye or data collection at the discretion of the Investigator and/or ophthalmologist.
6. Any corrected visual acuity < 20/20, or intraocular pressure ≥ 20 mmHg.
7. Subjects who wear contact lenses within 1 month prior to administration, or will wear contact lenses during the trial.
8. Use of any prescription drugs excluding hormonal contraception, herbal supplements, or nonprescription drugs, including oral anti-histamines (for seasonal allergies) or ophthalmology drugs, within 1 month (30 days) or 5 half-lives (whichever is longer) prior to study drug administration, or dietary supplements within 1 week prior to study drug administration, unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study. Over-the-counter multivitamins will be permitted. If needed, paracetamol/acetaminophen may be used, but must be documented in the concomitant medications/significant non-drug therapies page of the source data. Exclusion applies to the use of Tropicamide 1% for the dilated retinal examination during baseline and final visit. Any questions of concomitant medications should be directed to the Sponsor.
9. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
10. Donation of blood 12 week prior to dosing.
11. Pregnant, or nursing females.
12. A history of psychiatric and psychological condition that, in the judgment of the investigator, may interfere with the planned treatment and follow-up, affect subject compliance or place the subject at high risk from treatment-related complications
13. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTcF interval > 450 milliseconds [ms], Bazett Formula: QTc = QT/RR0.5）at Screening and on Day -1.
14. Active hepatitis B or C. HBV carriers without active disease (HBV DNA titer < 1000 cps/mL or 200 IU/mL), or cured Hepatitis C (negative HCV RNA test) may be enrolled, in the judgement of the investigator.
15. Human immunodeficiency virus (HIV) positive.
16. Immunization with a live or attenuated vaccine is prohibited within 4 weeks prior to study drug administration. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed)
17. History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]) or positive alcohol breath test at screening
18. History of significant drug abuse within one year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening
19. Positive urine drug screen, cotinine test, or alcohol breath test at screening
20. Any reason which, in the opinion of the Investigator and Monitor, would prevent the subject from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of AE reporting for safety and tolerability (SDE) | 31 days
  AEs are documented and recorded per Guidance for Industry Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials.
Incidence of SAE reporting for safety and tolerability (SDE) | through study completion, an average of 1 year
Body temperature for safety and tolerability (SDE) | 8 days for follow-up visit
Pulse rate for safety and tolerability (SDE) | 8 days for follow-up visit
Respiration rate for safety and tolerability (SDE) | 8 days for follow-up visit
Blood pressure for safety and tolerability (SDE) | 8 days for follow-up visit
Incidence of discomfort by clinical inquiring and observation for safety and tolerability (SDE) | 8 days for follow-up visit
Incidence of abnomal physical findings for safety and tolerability (SDE) | 8 days for follow-up visit
  Via physical examination. Full physical examination including the cardiovascular, pulmonary, gastrointestinal, and nerve system and skin will be performed at screening and end of study visits, and partial physical examination can be done to assess any abnormalities or change from baseline, including focused skin and cardiopulmonary examination, and as clinically indicated.
Visual acuity for safety and tolerability (SDE) | 8 days for follow-up visit
Intraocular pressure for safety and tolerability (SDE) | 8 days for follow-up visit
  Via tonopen or Goldmann tonometer.
Incidence of abnomal extraocular and anterior segament findings for safety and tolerability (SDE) | 8 days for follow-up visit
  Via bare eye and a slit lamp microscopy. Examination includes eyelid, cornea, anterior chamber, lens and conjunctiva (palpebral and bulbar).
  Fluorescein staining of cornea and conjunctival surfaces under a slit lamp microscopy.
White blood cell, red blood cell, platelet count, absolute neutrophils, monocytes , lymphocytes esoinophils and basophils (SDE) | 8 days for follow-up visit
  Unit: X10E3/uL. In hematology for safety and tolerability
Percentage of netrophils, monocytes, lymphocytes, eosinophils, basophils, hematocrit and mean cellular HGB concentration in hematology (SDE) | 8 days for follow-up visit
  Unit: %. In hematology for safety and tolerability
Mean cellulara HGB in hematology (SDE) | 8 days for follow-up visit
  Unit: pg. In hematology for safety and tolerability
Mean cellular volume in hematology (SDE) | 8 days for follow-up visit
  Unit: fL. In hematology for safety and tolerability
Hemoglobin in hematology (SDE) | 8 days for follow-up visit
  Unit: g/dL. In hematology for safety and tolerability
Weight (SDE) | 8 days for follow-up visit
  Unit: kg. In chemistry for GFP calculation
Akaline phosphatase, ALT, amylase, AST, creatine kinase, GGT and LDH in chemistry (SDE) | 8 days for follow-up visit
  Unit: U/L. In chemistry for safety and tolerability
Serum chloride, potassium and sodium in chemistry (SDE) | 8 days for follow-up visit
  Unit: mmol/L. In chemistry for safety and tolerability
Direct bilirubin, total bilirubin, urea nitrogen, calcium, cholesterol, creatinine, fasting glucose, triglycerides and uric acid in chemistry (SDE) | 8 days for follow-up visit
  Unit: mg/dL. In chemistry for safety and tolerability
GFR estimate (Cockcroft-Gault) in chemistry (SDE) | 8 days for follow-up visit
  Unit: mL/min. In chemistry for safety and tolerability
Albumin, globulin, total protein in chemistry (SDE) | 8 days for follow-up visit
  Unit: g/dL. In chemistry for safety and tolerability
A/G ratio in chemistry (SDE) | 8 days for follow-up visit
  Unit: NA. In chemistry for safety and tolerability
Partial thromboplastin time, prothrombin time and thrombin time in coagulation (SDE) | 8 days for follow-up visit
  Unit: second. Unit: second. In coagulation for safety and tolerability
Fibrinogen in coagulation (SDE) | 8 days for follow-up visit
  Unit: mg/dL. In coagulation for safety and tolerability
International normalized ratio in coagulation (SDE) | 8 days for follow-up visit
  Unit: NA In coagulation for safety and tolerability
Incidence of abnormal urine analysis by blood, glucose, ketones, leukocyte, protein, nitrite, bilirubin and urobilinogen in urine analysis (SDE) | 8 days for follow-up visit
  Unit: QUAL. In urine analysis for safety and tolerability
PH in urine analysis (SDE) | 8 days for follow-up visit
  Unit: NA In urine analysis for safety and tolerability
Specific gravity in urine analysis (SDE) | 8 days for follow-up visit
  Unit: NA In urine analysis for safety and tolerability
Heart rate for safety and tolerability (SDE) | 8 days for follow-up visit
  By triplicate 12-lead electrocardiogram
QRS wave interval, QT interval, QTC interval, PQ interval, P wave interval and RR interval for safety and tolerability (SDE) | 8 days for follow-up visit
  By triplicate 12-lead electrocardiogram
QRS angle value for safety and tolerability (SDE) | 8 days for follow-up visit
  By triplicate 12-lead electrocardiogram
QTCF value for safety and tolerability (SDE) | 8 days for follow-up visit
  By triplicate 12-lead electrocardiogram
Satisfaction assessed by Ocular Surface Disease Index (OSDI) questionnaires for safety and tolerability (SDE) | 8 days for follow-up visit
  0-100 points. Higher score means more severe discomfort of ocular surface.
Satisfaction assessed by National Eye Institute 25-Item Visual Function (NEI-VFQ25) questionnaires for safety and tolerability (SDE) | 8 days for follow-up visit
  0-100 points. Higher score means better vision function.
Incidence of AE reporting for safety and tolerability (RDE) | 48 days
  AEs are documented and recorded per Guidance for Industry Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials.
Incidence of SAE reporting for safety and tolerability (RDE) | Through study completion, an average of 1 year
Body temperature for safety and tolerability (RDE) | 15 days for follow-up visit
Pulse rate for safety and tolerability (RDE) | 15 days for follow-up visit
Respiration rate for safety and tolerability (RDE) | 15 days for follow-up visit
Blood pressure for safety and tolerability (RDE) | 15 days for follow-up visit
Incidence of discomfort by clinical inquiring and observation for safety and tolerability (RDE) | 15 days for follow-up visit
Incidence of abnomal physical findings for safety and tolerability (RDE) | 15 days for follow-up visit
  Via physical examination. Full physical examination including the cardiovascular, pulmonary, gastrointestinal, and nerve system and skin will be performed at screening and end of study visits, and partial physical examination can be done to assess any abnormalities or change from baseline, including focused skin and cardiopulmonary examination, and as clinically indicated.
Visual acuity for safety and tolerability (RDE) | 15 days for follow-up visit
Intraocular pressure for safety and tolerability (RDE) | 15 days for follow-up visit
  Via tonopen or Goldmann tonometer.
Incidence of abnomal extraocular and anterior segament findings for safety and tolerability (RDE) | 15 days for follow-up visit
  Via bare eye and a slit lamp microscopy. Examination includes eyelid, cornea, anterior chamber, lens and conjunctiva (palpebral and bulbar).
  Fluorescein staining of cornea and conjunctival surfaces under a slit lamp microscopy.
Incidence of abnormal findings from dilated fundus exam (RDE) | 15 days for follow-up visit
  Dilated fundus exam for once at D15.
White blood cell, red blood cell, platelet count, absolute neutrophils, monocytes , lymphocytes esoinophils and basophils in hematology for safety and tolerability (RDE) | 15 days for follow-up visit
  Unit: X10E3/uL. In hematology for safety and tolerability
Percentage of netrophils, monocytes, lymphocytes, eosinophils, basophils, hematocrit and mean cellular HGB CON/MCHC in hematology (RDE) | 15 days for follow-up visit
  Unit: %. In hematology for safety and tolerability
Mean cellulara HGB in hematology (RDE) | 15 days for follow-up visit
  Unit: pg. In hematology for safety and tolerability
Mean cellular volume in hematology (RDE) | 15 days for follow-up visit
  Unit: fL. In hematology for safety and tolerability
Hemoglobin in hematology (RDE) | 15 days for follow-up visit
  Unit: g/dL . In hematology for safety and tolerability
Weight (RDE) | 15 days for follow-up visit
  Unit: kg. In chemistry for GFP calculation
Akaline phosphatase, ALT, amylase, AST, creatine kinase, GGT and LDH in chemistry (RDE) | 15 days for follow-up visit
  Unit: U/L. In chemistry for safety and tolerability
Serum chloride, potassium and sodium in chemistry (RDE) | 15 days for follow-up visit
  Unit: mmol/L. In chemistry for safety and tolerability
Direct bilirubin, total bilirubin, urea nitrogen, calcium, cholesterol, creatinine, fasting glucose, triglycerides and uric acid in chemistry (RDE) | 15 days for follow-up visit
  Unit: mg/dL. In chemistry for safety and tolerability
GFR estimate (Cockcroft-Gault) in chemistry (RDE) | 15 days for follow-up visit
  Unit: mL/min. In chemistry for safety and tolerability
Albumin, globulin, total protein in chemistry (RDE) | 15 days for follow-up visit
  Unit: g/dL. In chemistry for safety and tolerability
A/G ratio in chemistry (RDE) | 15 days for follow-up visit
  Unit: NA. In chemistry for safety and tolerability
Partial thromboplastin time, prothrombin time and thrombin time in chemistry (RDE) | 15 days for follow-up visit
  Unit: second. In coagulation for safety and tolerability
Fibrinogen in coagulation (RDE) | 15 days for follow-up visit
  Unit: mg/dL. In coagulation for safety and tolerability
International normalized ratio in coagulation (RDE) | 15 days for follow-up visit
  Unit: NA. In coagulation for safety and tolerability
Incidence of abnormal urine analysis by blood, glucose, ketones, leukocyte, protein, nitrite, bilirubin and urobilinogen in urine analysis (RDE) | 15 days for follow-up visit
  Unit: QUAL. In urine analysis for safety and tolerability
PH in urine analysis (RDE) | 15 days for follow-up visit
  Unit: NA. In urine analysis for safety and tolerability
Specific gravity in urine analysis (RDE) | 15 days for follow-up visit
  Unit: NA. In urine analysis for safety and tolerability
Heart rate for safety and tolerability (RDE) | 15 days for follow-up visit
  By triplicate 12-lead electrocardiogram
QRS wave interval, QT interval, QTC interval, PQ interval, P wave interval and RR interval for safety and tolerability (RDE) | 15 days for follow-up visit
  By triplicate 12-lead electrocardiogram
QRS angle value for safety and tolerability (RDE) | 15 days for follow-up visit
  By triplicate 12-lead electrocardiogram
QTCF value for safety and tolerability (RDE) | 15 days for follow-up visit
  By triplicate 12-lead electrocardiogram
Satisfaction assessed by Ocular Surface Disease Index (OSDI) questionnaires for safety and tolerability (RDE) | 15 days for follow-up visit
  0-100 points. Higher score means more severe discomfort of ocular surface.
Satisfaction assessed by National Eye Institute 25-Item Visual Function (NEI-VFQ25) questionnaires for safety and tolerability (RDE) | 15 days for follow-up visit
  0-100 points. Higher score means better vision function.

SECONDARY OUTCOMES:
AUC0-∞ in each SDE cohort | 2 days
AUC0-t in each SDE cohort | 2 days
Cmax in each SDE cohort | 2 days
t1/2 in each SDE cohort | 2 days
CL in each SDE cohort | 2 days
Vd in each SDE cohort | 2 days
AUC0-∞ in each RDE cohort | 8 days
AUC0-t in each RDE cohort | 8 days
Cmax in each RDE cohort | 8 days
t1/2 in each RDE cohort | 8 days
CL in each RDE cohort | 8 days
Vd in each RDE cohort | 8 days

OTHER OUTCOMES:
Alcohol breath test (SDE) | 8 days for follow-up visit
Urine drug screening (SDE) | 8 days for follow-up visit
  Urine drug screening includes amphetamine, barbiturates, benzodiazepines, buprenorphine/metabolite, cocaine, cotinine, opiates, oxycodone, PCP, MDMA, methadone, methamphetamine, THC and tricyclic antidepressants.
Serum pregnancy test for females (SDE) | 8 days for follow-up visit
Alcohol breath test (RDE) | 15 days for follow-up visit
Urine drug screening (RDE) | 15 days for follow-up visit
  Urine drug screening includes amphetamine, barbiturates, benzodiazepines, buprenorphine/metabolite, cocaine, cotinine, opiates, oxycodone, PCP, MDMA, methadone, methamphetamine, THC and tricyclic antidepressants.
Serum pregnancy test for females (RDE) | 15 days for follow-up visit

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel International, Glendale, California, United States